CLINICAL TRIAL: NCT04690660
Title: Swiss Postpartum Hypertension Cohort (Swiss-PPHT)
Brief Title: Swiss Postpartum Hypertension Cohort
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00736; me20Burkard
Record Dates: First submitted 2020-12-15; First posted 2020-12-31 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Hypertension (PPHT)
Keywords: Pregnancy Induced Hypertension (PIH); Home Blood Pressure Monitoring (HBPM); Office Blood Pressure Monitoring (OBPM); Automated Office Blood Pressure Measurement (AOBPM); Gestational Hypertension; HekaHealth Self-Measured Blood Pressure (SMBP) App
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Alzheimer Disease | interventions — Data Collection; Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for biomarker
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection for parameters of organ damage (cardiac and renal blood markers) — Blood results will be taken out of next routine venipuncture. Routinely collected standard parameters are a blood count, chemistry panel including renal parameters and electrolytes, lipid profile and a HbA1c as well as albumin/creatinine and protein/creatinine ratio in urine.
Other: Data collection for blood pressure (BP) — Clinic blood pressure and 24hour BP Measurements
Other: Home-based blood pressure management (substudy) — Subjects participating in home-based blood pressure management via telemonitoring will receive a free HekaHealth application (App) for the structured assessment of HBPM.
Other: Biomarker Profiles (substudy) — Substudy where possible cardiac, renal and pregnancy related biomarkers will be additionally analyzed. The following biomarkers will be analyzed: N terminal (NT)-proBNP, Troponin, elevated mid-regional pro-atrial natriuretic peptide (ANP), elevated mid-regional pro adrenomedullin (ADM), soluble fms-like tyrosine kinase (sFlt-1), and placenta growth factor (PlGF).
Other: Data collection on patient reported outcomes — Data collection on patient reported outcomes (Questionnaire EQ-5D, Questionnaire for App based monitoring )

SUMMARY:
This open label, prospective observational, single-center registry is to study short-, intermediate-and long-term course of postpartum hypertension and predictors/risk factors associated with long term cardiovascular and renal risk.

Current disease management strategies will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* all women with hypertensive disorders of pregnancy
* postpartum hypertension (blood pressure measurements of systolic ≥140 and/or diastolic ≥ 90mmHg or antihypertensive therapy within the first 14 days after delivery)
* women with preexisting hypertension or
* women on antihypertensive medication

Exclusion Criteria:

* delivery > 14 days
* lack of consent to participate in the study, language barriers or lack of general understanding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will take place at the Hypertension Clinic of the Medical Outpatient Department at the University Hospital Basel and the Department of Obstetrics and Gynaecology at the University Hospital Basel. Participants will be consecutively screened and recruited by the treating physicians and the Hypertension Team of the Hypertension Clinic.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of persistent hypertension defined by 24 hours BP measurement | through study completion, an average of 5 years
  Frequency of persistent hypertension defined by 24 hours BP measurement
Frequency of persistent hypertension defined by office blood pressure measurement (OBPM, AOBPM) | through study completion, an average of 5 years
  Frequency of persistent hypertension defined by office blood pressure measurement (OBPM, AOBPM)
Frequency of microalbuminuria | through study completion, an average of 5 years
  Frequency of microalbuminuria
Frequency of damage to the retina of the eyes (retinopathy) | through study completion, an average of 5 years
  Frequency of damage to the retina of the eyes (retinopathy)
Signs of hypertensive heart disease | up to 24 months
  Signs of hypertensive heart disease at transthoracic echocardiography determined by left ventricular hypertrophy (LVH)
Frequency of dyslipidemia | through study completion, an average of 5 years
  Frequency of dyslipidemia
Frequency of prediabetes/diabetes | through study completion, an average of 5 years
  Frequency of prediabetes/diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Thenral Socrates, Dr. med., Principal Investigator — Medical Outpatient Department and Hypertension Clinic, University Hospital BaselUni
Locations (1):
- Medical Outpatient Department and Hypertension Clinic, University Hospital Basel, Basel, Switzerland